CLINICAL TRIAL: NCT04118907
Title: Effects of Sound Stimulation, Somatosensory Stimulation, Vestibular Stimulation and the Combinations on Tinnitus Loudness and Tinnitus Related Distress in Patients
Brief Title: Different Stimuli Were Given to Patients With Chronic Pure Tone Tinnitus to Verify the Effective Treatment of Tinnitus.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dan Su (Other)
Responsible Party: Sponsor-Investigator, Dan Su, principal investigator, The First Affiliated Hospital of Anhui Medical University
Organization: The First Affiliated Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mssftinnitus
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Tinnitus; Acoustic Stimulation; Somatic Stimulation; Vestibular Stimulation
Keywords: tinnitus; stimulation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- acoustic stimulation (Experimental): Pink noise in both ears is given to tinnitus patients. The pink noise is removed by notch filter from tinnitus frequencies that are 20 decibel higher than the threshold.
  Interventions: Device: multiple sensory stimulation
- somatic stimulation (Experimental): Three stimulation points were selected for each ear of tinnitus patients, namely ear door (CN.V), auditory Palace (CN.VII) and Yifeng (C2/3). The stimulation intensity should be needle-sensed.
  Interventions: Device: multiple sensory stimulation
- vestibular stimulation (Experimental): The patient sat on a rotating chair with sinusoidal harmonic acceleration and rotated without causing the greatest frequency of discomfort.
  Interventions: Device: multiple sensory stimulation
- acoustic + somatic stimulation (Experimental): Combination of auditory and somatic stimulation for tinnitus patients
  Interventions: Device: multiple sensory stimulation
- acoustic + vestibular stimulation (Experimental): Combination of auditory and vestibular stimulation for tinnitus patients
  Interventions: Device: multiple sensory stimulation
- acoustic + somatic + vestibular stimulation (Experimental): Combination of auditory stimulation, somatic stimulation and vestibular stimulation for tinnitus patients
  Interventions: Device: multiple sensory stimulation

INTERVENTIONS:
Device: multiple sensory stimulation — The patients were recruited to record their medical history, and the hearing level, tinnitus indicators, vestibular function and tinnitus disability indicators were tested. Then the patients were randomly divided into six groups. They received the corresponding stimulation 20 minutes a day, 5 days a week for 3 weeks. After the last stimulation, the above tests were repeated immediately, one week later and three months later.

SUMMARY:
In this experiment, patients with chronic pure tone tinnitus were divided into three groups to receive auditory stimulation, somatosensory stimulation, vestibular stimulation and combined stimulation, in order to find an effective way to treat tinnitus

DETAILED DESCRIPTION:
120 patients with chronic pure tone tinnitus over 6 months were randomly divided into 6 groups, one group was given auditory stimulation, one group was given somatosensory stimulation, one group was given auditory stimulation + somatosensory stimulation, one group was given auditory stimulation + vestibular stimulation, the last group was given auditory stimulation + somatosensory stimulation + vestibular stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Pure tone tinnitus
* Unilateral and bilateral
* female and male
* Tinnitus has a history of more than 6 months

Exclusion Criteria:

* Pulsatile tinnitus of blood vessel
* Meniere's disease
* Chronic headache
* Neurological diseases (such as brain tumors)
* Patients with mental / mental illness undergoing treatment
* Pregnant women and patients with other untreatable diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Electrical audiometry and acoustic impedance | Three months from the time the patient was selected to the end of the stimulus
  Assessment of hearing in patients
Tinnitus frequency and loudness | Three months from the time the patient was selected to the end of the stimulus
  Detection of tinnitus frequency and loudness in patients
Tinnitus disability scale | Three months from the time the patient was selected to the end of the stimulus
  Tinnitus handicap inventory score was used to detect the degree of tinnitus.0-16 points without disability, 18-36 points with mild disability, 38-56 points with moderate disability and 58-100 points with severe disability. The 95% confidence interval is 20 points, that is, the difference between the two tests before and after the experiment is greater than or equal to 20 points.

CONTACTS AND LOCATIONS:
Overall Officials: Busheng Tong, doctor, Study Director — E.N.T. department of the First Affiliated hospital of Anhui Medical University
Locations (1):
- E.N.T. department of the First Affiliated hospital of Anhui Medical University, Hefei, Anhui, China